CLINICAL TRIAL: NCT07038369
Title: A Phase 1 Study of a Selective AKT1 E17K Allosteric Inhibitor, ATV-1601, in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of ATV-1601 in Patients With Advanced Cancer That Have AKT1 E17K Mutations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atavistik Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATV-1601-101
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors; Breast Cancer; Breast Carcinoma; Breast Neoplasms; ER Positive Breast Cancer; Cervical Cancers; Cervical Neoplasms; Cervical Carcinoma; Triple Negative Breast Cancer; Gynecologic Cancers; Gynecologic Neoplasm; Endometrial Cancer; Endometrial Neoplasm; Endometrial Carcinoma (EC); Fallopian Cancer; Ovarian Carcinoma; Ovarian Cancer; Ovarian Neoplasms; Prostate Cancers; Prostate Carcinoma; Solid Tumors; Neoplasms; Neoplasms by Site; Breast Diseases; Uterine Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms
Keywords: AKT mutation; Mutant AKT; AKT1 mutation; AKT mutant; Gynecologic carcinoma; Fallopian Carcinoma; Fallopian Neoplasm; HR positive breast; AKT Gene Mutation; AKT1 E17K
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Triple Negative Breast Neoplasms; Genital Neoplasms, Female; Endometrial Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Neoplasms; Neoplasms by Site; Breast Diseases; Uterine Neoplasms; Urogenital Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental/Part 1a: ATV-1601 (Experimental): ATV-1601
  Interventions: Drug: ATV-1601
- Experimental/Part 1b: ATV-1601 + Fulvestrant (Experimental): ATV-1601 + Fulvestrant
  Interventions: Combination Product: ATV-1601 + Fulvestrant

INTERVENTIONS:
Drug: ATV-1601 — Drug: ATV-1601
  • Oral ATV-1601
  Arms: Experimental/Part 1a: ATV-1601
Combination Product: ATV-1601 + Fulvestrant — Drug: ATV-1601
  * Oral ATV-1601 Drug: Fulvestrant
  * Intramuscular Injection
  Arms: Experimental/Part 1b: ATV-1601 + Fulvestrant

SUMMARY:
This is a Phase 1, open-label study to evaluate the safety and tolerability of ATV-1601 administered orally in adults with AKT1 E17K-mutant, advanced solid tumors and also in HR+/HER2- advanced and metastatic breast cancer, with or without fulvestrant.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, multicenter, Phase 1a/1b dose escalation dose finding, and dose expansion study to evaluate safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of ATV-1601 as monotherapy in participants with advanced or metastatic solid tumors with the AKT1 E17K mutation, and in combination with fulvestrant in participants with breast cancer that has the AKT1 E17K mutation. This study has a dose escalation and expansion phase with ATV-1601, and an escalation and expansion phase in combination with Fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic or advanced-stage solid malignant tumor or HR+/HER2- breast cancer.
2. Have progressed on, were intolerant to, or experienced disease recurrence after standard therapy and have no available effective or tolerable treatment options to derive clinically meaningful benefit.
3. Tumor must have documented specific mutation profile as outlined below based on local laboratory testing.
4. Participants with solid tumors or HR+/HER2- breast cancer with AKT1 E17K mutations.
5. Measurable disease according to RECIST v1.1 criteria.
6. Formalin-fixed paraffin-embedded tumor specimen available for submission.
7. Eastern Cooperative Oncology Group performance status of 0 or 1.

Exclusion Criteria:

1. Previously documented activating mutations in KRAS, NRAS, HRAS, or BRAF.
2. Inadequate bone marrow reserve or organ function.
3. Clinically significant abnormalities of glucose metabolism.
4. Participants who are symptomatic or have uncontrolled brain metastases.
5. Requires treatment with certain medications.

Participants must meet other inclusion/exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Expansion: Maximum and minimum plasma concentration | Approximately 48 months.
  Drug concentration in Blood.
Expansion: Time to C Max | Approximately 48 months
  Drug concentration in Blood
Expansion: Area under the concentration-time curve | Approximately 48 months
  Drug concentration in Blood
Expansion: AUC at end of dosing interval | Approximately 48 months
  Drug concentration in Blood
Expansion: AUC extrapolated to infinity | Approximately 48 months
  Drug concentration in Blood
Expansion: Half-life | Approximately 48 months
  Drug concentration in Blood
Expansion: Trough Concentrations | Approximately 48 months
  Drug concentration in Blood
Escalation & Expansion: Safety and Tolerability of monotherapy. | Approximately 48 months.
  Number of participants with Treatment Emergent Adverse Events (TEAEs). Safety will be assessed by monitoring adverse events, laboratory tests and ECG results.
Escalation: Maximum tolerated dose and/or recommended phase 2 dose of ATV-1601 in monotherapy. | Approximately 48 months.
  Number of patients with dose-limiting toxicities.
Escalation: Maximum tolerated dose and/or recommended phase 2 dose of ATV-1601 combination with fulvestrant. | Approximately 48 months.
  Number of patients with dose-limiting toxicities.

SECONDARY OUTCOMES:
Escalation: Maximum and minimum plasma concentration | Approximately 48 months.
  Drug concentration in Blood.
Escalation: Time to C max | Approximately 48 months
  Drug concentration in Blood
Escalation: Area under the concentration-time curve | Approximately 48 months
  Drug concentration in Blood
Escalation: AUC at end of dosing interval | Approximately 48 months
  Drug concentration in Blood
Escalation: AUC extrapolated to infinity | Approximately 48 months
  Drug concentration in Blood
Escalation: Half-life | Approximately 48 months
  Drug concentration in Blood
Escalation: Trough Concentrations | Approximately 48 months
  Drug concentration in Blood
Escalation & Expansion: Objective response rate | Approximately 48 months
  Tumor measurements by RECIST 1.1
Escalation & Expansion: Duration of Response | Approximately 48 months
  Tumor measurements by RECIST 1.1
Escalation & Expansion: Clinical Benefit Rate | Approximately 48 months
  Tumor measurements by RECIST 1.1
Expansion: Progression Free Survival | Approximately 48 months
  Tumor measurements by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Atavistik Bio
Locations (13):
- United States (8):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Florida Cancer Specialists & Research Institute - Lake Mary, Lake Mary, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
- Centre Leon Berard, Lyon, France
- National Cancer Centre Singapore, Singapore, Singapore
- Spain (3):
  - Hospital Clinic Barcelona, Barcelona
  - START Madrid - Hospital Fundacion Jimenez Diaz, Madrid
  - START Madrid - CIOCC, Madrid